CLINICAL TRIAL: NCT01670851
Title: Perineal Reconstruction Following Extralevator Abdominoperineal Excision of Rectum and Simultaneous Stoma Sublay Reinforcement
Brief Title: Perineal Reconstruction Following eLAPE and Simultaneous Stoma Sublay Reinforcement
Acronym: PRESSUR
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Karolinska University Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Slagelse Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ISIS.11.01.06.BS/SC
Record Dates: First submitted 2012-08-19; First posted 2012-08-22 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Rectal Cancer
Keywords: eLAPE,; perineum,; pelvic floor reconstruction
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Strattice: eLAPE
  Interventions: Device: Strattice

INTERVENTIONS:
Device: Strattice — Perineal reconstruction and stoma reinforcement with Strattice

SUMMARY:
This is a prospective, multicenter, single arm, observational pilot study to assess the clinical outcomes of Strattice Reconstructive Tissue Matrix for perineal reconstruction following eLAPE and simultaneous stoma reinforcement.

DETAILED DESCRIPTION:
About 40 subjects will be enrolled from 4 centers over approx 24 months. Subjects will all be undergoing extralevator abdominoperineal excision with concomitant ostomy creation.

ELIGIBILITY:
Inclusion Criteria:

* Primary cancers undergoing curative surgery (R0)
* Life expectancy > 2 yrs
* Neoadjuvant radiotherapy with or without chemotherapy

Exclusion Criteria:

* Pelvic extenteration or extended resections
* Previously irradiated patients (i.e. radiation therapy for a previous cancer)
* Co-morbidities of: systemic infection, chronic liver failure, chronic renal failure, HIV, Hepatitis C, other advanced/metastatic cancer, collagen disorder
* sensitivity to porcine derived products or polysorbate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with low rectal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Perineal wound healing | 12 months
  Perineal wound healing will be assessed using the Southamptom Wound Scoring System and perineal pain assessed using a visual analogue scale (VAS) daily during hospital stay and then POD 7, 30 and months 3, 6 and 12.

SECONDARY OUTCOMES:
Incidence of perineal herniation | 24 months
  Incidence of perineal hernia
Incidence of parastomal hernia | 24 months
  Stoma will be assessed for herniation at Months 3, 6, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Baljit Singh, FRCS, FACS, Principal Investigator — University Hospital Leicester, UK; Sanjay Chaudhri, FRCS, Principal Investigator — University Hospital Leicester, UK; Per J Nilsson, MD, Principal Investigator — Karolinska Institutet; Pierre J Maina, MD, Principal Investigator — Slagelse Hospital, Denmark; W Bemelman, MD, Principal Investigator — Academic Medical Center, Amsterdam, Netherlands
Locations (3):
- Slagelse Hospital, Slagelse, Denmark
- Karolinska University Hospital, Stockholm, Sweden
- University Hospitals Leicester, Leicester, United Kingdom